CLINICAL TRIAL: NCT01691378
Title: Window to Hope-Evaluating a Psychological Treatment for Hopelessness Among Veterans With Traumatic Brain Injury
Acronym: WtoH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Brenner (U.S. Federal Agency)
Collaborators: Military Suicide Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Lisa Brenner, Psychologist, MIRECC Director, VA Eastern Colorado Health Care System
Organization: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0127
Record Dates: First submitted 2012-06-05; First posted 2012-09-24 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Traumatic Brain Injury; Hopelessness; Suicide
Keywords: Veterans; Window to Hope; Cognitive Behavioral Therapy; Traumatic Brain Injury; Hopelessness; Suicide
MeSH Terms: conditions — Brain Injuries, Traumatic; Suicide

STUDY DESIGN:
Intervention Model Description: After enrollment, participants were randomized to either receive the WtoH Intervention first, or Waitlist Control. After Time 2, the Waitlist Control arm crosses over and has the opportunity to participate in the WtoH Intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- WtoH Intervention (Experimental): Window to Hope: Psychotherapy consists of 10 2-hour sessions for a maximum dose delivered of 20 hours. Therapy consists of small groups of up to 2 participants.
  Interventions: Other: Window to Hope
- Waitlist Control (Other): Members of the Waitlist Control arm continued to receive nonconstrained usual care from the Veterans Health Administration. Those initially allocated to the Waitlist Control arm were later provided with the opportunity to cross over and receive the WtoH Intervention after Time 2.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Other: Window to Hope — Psychotherapy - Group
  Arms: WtoH Intervention
Other: Waitlist Control — Members of the Waitlist Control arm continued to receive nonconstrained usual care from the Veterans Health Administration. Those initially allocated to the Waitlist Control arm were later provided with the opportunity to cross over and receive the WtoH Intervention after Time 2.
  Arms: Waitlist Control

SUMMARY:
The purpose of this project is to provide further evidence regarding a groundbreaking psychological treatment for suicide prevention in individuals with moderate to severe traumatic brain injury (TBI), Window to Hope (WtoH). The study will be one of the first five randomized clinical trials (RCTs) internationally to evaluate a psychological treatment for affective distress after TBI and the first conducted in the United States (U.S.) to specifically address suicide risk as an outcome.

The current project aims to adapt WtoH for U.S. military personnel/Veterans (expert Consensus Conference, participant total up to 15), implement the intervention in a Veterans Affairs Medical Center (VAMC) (Pilot Groups 1-4, participant total up to 12), and replicate the results from the original trial in this novel context with a larger sample size (n=70 completed protocols [up to 90 recruited]. Deliverables are expected to include an intervention suitable for both dissemination and larger Phase III trials.

DETAILED DESCRIPTION:
Prior to implementing the intervention, Dr. Simpson will work with VA study team members (e.g., Drs. Brenner, Matarazzo, Signoracci) to modify WtoH manual semantics and graphics to meet the needs of the U.S. Veteran population. Dr. Brenner has a long history of working within the Veterans Health Administration (VHA) and is a Diplomate in Rehabilitation Psychology. An expert committee (up to 15 participants) will also be convened for a meeting focused on the cross-cultural adaptation of WtoH. All efforts will be made to include experts in treating TBI and stakeholders (e.g., Veterans with or without TBI and/or family members/support persons) on the committee. Members of the research team will contact potential committee members by phone, email, mail or in person. Presentations may also be made to Veterans/family members/support persons receiving care, participating in patient advocacy activities, or providing peer support. Prior to reviewing the content, the expert committee will be provided background on the current state of knowledge about suicidality and hopelessness after TBI, available treatment options, and information regarding the underlying theoretical basis and key features of the WtoH program. The committee will then review the ten sessions to identify potential changes required to the therapeutic content, exercises, language and graphics to ensure that it is culturally appropriate for the VAMC context. Modifications will be made employing a consensus approach among the expert committee.

The adapted program will then be trialed across four pilot groups. Once the pilot groups have been completed (see below) the expert committee will be reconvened for a final review of the program. Data collected on acceptability and feasibility will be presented to the committee and test therapists. Any necessary final modifications to assessment procedures and/or the intervention to ensure that the program is appropriate for the Veterans' condition will be made employing a consensus approach.

The revised version of the manual will be used to conduct the RCT. Up to 90 Veterans will participate.

ELIGIBILITY:
Inclusion Criteria for Pilot Groups:

* Age between 18 and 89
* Determination of positive history of moderate/or severe TBI
* Ability to adequately respond to questions regarding the informed consent procedure

Exclusion Criteria for Pilot Groups:

* History of alcohol abuse in the seven days prior to baseline assessment
* History of non-alcohol substance abuse within the last 30 days prior to baseline assessment
* Same-day drug or alcohol abuse during treatment
* History of mild TBI only
* Inability to travel to the Denver VA for daily or weekly therapy sessions

Inclusion Criteria for RCT:

* Age between 18 and 65
* Determination of positive history of moderate/or severe TBI
* Beck Hopelessness Scale score of 9 or greater
* Ability to adequately respond to questions regarding the informed consent procedure

Exclusion Criteria for RCT:

* Diagnosis of neurological condition(s)
* History of alcohol abuse in the seven days prior to baseline assessment
* History of non-alcohol substance abuse within the last 30 days prior to baseline assessment
* Same-day drug or alcohol abuse during treatment
* History of mild TBI only
* Inability to travel to the Denver VA for weekly therapy sessions

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2015-10-27 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, Ph.D., Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- VA Eastern Colorado Health Care System, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brenner LA, Forster JE, Hoffberg AS, Matarazzo BB, Hostetter TA, Signoracci G, Simpson GK. Window to Hope: A Randomized Controlled Trial of a Psychological Intervention for the Treatment of Hopelessness Among Veterans With Moderate to Severe Traumatic Brain Injury. J Head Trauma Rehabil. 2018 Mar/Apr;33(2):E64-E73. doi: 10.1097/HTR.0000000000000351. PMID 29084101
- [Background] Matarazzo BB, Hoffberg AS, Clemans TA, Signoracci GM, Simpson GK, Brenner LA. Cross-cultural adaptation of the Window to Hope: a psychological intervention to reduce hopelessness among U.S. veterans with traumatic brain injury. Brain Inj. 2014;28(10):1238-47. doi: 10.3109/02699052.2014.916419. Epub 2014 Jun 19. PMID 24946053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant issues
Groups:
- Waitlist Control: Participants in the Waitlist Control arm continued to receive nonconstrained usual care from the Veterans Health Administration. Waitlist Control arm participants were provided with the opportunity to cross over and receive the WtoH Intervention after Time 2 assessment, 3 months after Time 1 baseline.
Period: Overall Study
Arm/Group | WtoH Intervention | Waitlist Control
Started | 22 | 22
Completed | 15 | 20
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Population: Of the 44 baseline participants enrolled/randomized, 35 completed the Time 2 assessment and were analyzed.
Groups:
- Waitlist Control: Participants in the Waitlist Control arm continued to receive nonconstrained usual care from the Veterans Health Administration. Waitlist Control arm participants were provided with the opportunity to cross over and receive the WtoH Intervention after Time 2 assessment, 3 months after Time 1 baseline.
  Waitlist Control arm baseline values reported from the Time 1 assessment
- Total: Total of all reporting groups
Arm/Group | WtoH Intervention | Waitlist Control | Total
Number analyzed (Participants) | 15 | 20 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 20 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.1) | 54.6 (8.8) | 51.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 13 | 19 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 15 | 20 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 10 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 20 | 35
Beck Hopelessness Scale [Mean (Standard Deviation); unit: units on a scale] — The Beck Hopelessness Scale (BHS) is a 20-item true/false self-report scale that measures negative expectations about the future held by respondents in the previous week. Scores range from 0 to 20, representing minimal (0-3), mild (4-8), moderate (9-14), and severe (>14) levels of hopelessness.
  units on a scale | 16.2 (3.2) | 14 (3.1) | 14.9 (3.3)
Beck Suicide Ideation Scale [Mean (Standard Deviation); unit: units on a scale] — The Beck Scale for Suicide Ideation (BSS) is a 19-item scale that assesses severity of suicidal ideation within the previous week, with total scores ranging from 0 (no suicidal ideation) to 38. Population: n=14 WtoH and n=19 Waitlist analyzed at Time 1 baseline due to incomplete BSS data for n=2 participants
  units on a scale
    number analyzed (Participants) | 14 | 19 | 33
    (all) | 5.0 (5.8) | 4.8 (5.5) | 4.91 (5.6)
Beck Depression Inventory-Second Edition [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory-Second Edition (BDI-II) is a self-report instrument measuring the severity of common depressive symptoms. Each of its 21 items is rated on a 4-point Likert scale ranging from 0 to 3; total scores range from 0 to 63, with higher scores indicating greater degrees of depressive symptomatology.
  units on a scale | 37.6 (11.6) | 28.4 (8.4) | 32.3 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Beck Hopelessness Scale (BHS)
Description: The BHS is a 20-item true-false self-report scale that measures the level of negative expectations about the future held by respondents over the previous week. Scores range from 0 to 20 representing nil (0-3), mild (4-8), moderate (9-14), and severe (>14) levels of hopelessness. Beck et al. found that BHS scores equal to or greater than 9 were associated with significantly elevated levels of suicide risk (Beck et al., 1985). As such, to be eligible to participate in this treatment trial individuals must have a score of 9 on the BHS at the time of screening and at the Time 1 baseline assessment. BHS outcome administered at the following study timepoints: Time 1 (Baseline for both arms), Time 2 (Post-Intervention for WtoH Intervention arm and Baseline 2 for Waitlist Control arm), and Time 3 Assessment (3 month follow up for WtoH Intervention arm and Post-Intervention for Waitlist Control arm.
Time Frame: Time 2 BHS was assessed 3-months after Time 1 baseline assessment for both arms of the trial. Time 3 BHS was assessed 6 months after Time 1 baseline for both arms of the trial.
Population: Participants were included in the outcome analysis if they completed the Time 2 assessment. N=14 participants from the WtoH Intervention first arm and n=16 participants from the Waitlist Control arm were analyzed at Time 3 due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Waitlist Control: Participants in the Waitlist Control arm continued to receive nonconstrained usual care from the Veterans Health Administration. Waitlist Control arm participants were provided with the opportunity to cross over and receive the WtoH Intervention after Time 2 assessment.
Arm/Group | WtoH Intervention | Waitlist Control
Number analyzed (Participants) | 15 | 20
score on a scale
  Time 2 BHS | 9.2 (5.6) | 12.6 (5.2)
  Time 3 BHS: number analyzed (Participants) | 14 | 16
  Time 3 BHS | 9.8 (5.6) | 8.9 (6.9)
Statistical Analysis 1: Comparison: WtoH Intervention vs Waitlist Control; Analyses 2-sided test w/ sig level .05. N=35 analyzed w/ α .05 provided 80% power to detect effect size d=1. T1 variables compared using Wilcoxon rank sum & Fisher exact tests. Per protocol analysis, all participants required T2 BHS. T2 BHS compared bet arms controlling for T1 BHS. No confounders significant at .10, not included in model. Analysis of covariance modeled T2 BHS as function of arm & T1 BHS. Estimated mean difference in T2 scores calculated, no adjustment for multiple comparisons; Test type: Superiority; p = .03, ANCOVA; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [.52 to 8.3]
Statistical Analysis 2: Comparison: Waitlist Control; Analysis contrasted T1 to T2 change with T2 to T3 change in Waitlist arm only. Waitlist participants serve as their own control & only variable controlled for was change in Waitlist period (if participants improved greatly during Waitlist period, they would no longer have enough "room" to change in Intervention period). Linear regression used with difference in change as dependent variable & Waitlist period change as only predictor. Estimated mean difference in change calculated from this model; Test type: Superiority; p = .01, Regression, Linear; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-7.9 to -1.3]
Statistical Analysis 3: Comparison: WtoH Intervention; Analysis investigated change from T1 to T3 within the WtoH Intervention first arm only. This difference was calculated and a 1-sample t test was used to determine whether the estimate was different from zero. As this change was not compared with a control group change, baseline values were not accounted for; Test type: Superiority; p = .0007, one-sample t-test; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-9.3 to -3.2]

2. Secondary Outcome: Beck Scale for Suicidal Ideation (BSS)
Description: The BSS is a 19-item scale that assesses severity of suicide ideation within the previous week with total scores ranging from 0 (no suicide ideation) to 38. High levels of internal consistency (Cronbach's α = .93) and concurrent validity have been reported with the Beck Depression Inventory (r =.64 to r =.75, Beck & Steer, 1993) as well as the BHS in Traumatic Brain Injury (TBI) (r =.60, Simpson & Tate, 2002) and non-brain-damaged populations (r =.52 to r = .63, Beck & Steer, 1993). BSS outcome administered at the following study timepoints: Time 1 (Baseline for both arms), Time 2 (Post-Intervention for WtoH Intervention arm and Baseline 2 for Waitlist Control arm), and Time 3 Assessment (3 month follow up for WtoH Intervention arm and Post-Intervention for Waitlist Control arm
Time Frame: Time 2 BSS was assessed 3-months after Time 1 baseline assessment for both arms of the trial. Time 3 BSS was assessed 6 months after Time 1 baseline for both arms of the trial.
Population: n=14 WtoH and n=19 Waitlist analyzed at Time 2 assessment due to incomplete BSS data for n=2 participants; n=13 WtoH and n=15 Waitlist BSS analyzed at Time 3 due to loss to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WtoH Intervention | Waitlist Control
Number analyzed (Participants) | 15 | 20
score on a scale
  Time 2 BSS: number analyzed (Participants) | 14 | 19
  Time 2 BSS | 2.0 (3.9) | 5.8 (6.9)
  Time 3 BSS: number analyzed (Participants) | 13 | 15
  Time 3 BSS | 1.9 (3.7) | 4.9 (7.3)
Statistical Analysis 1: Comparison: WtoH Intervention vs Waitlist Control; Analyses 2-sided test w/ sig level .05. N=35 analyzed w/ α .05 provided 80% power to detect effect size d=1. T1 variables compared using Wilcoxon rank sum & Fisher exact tests. Per protocol analysis, all participants required T2 BHS. T2 BSS compared bet arms controlling for T1 BSS. No confounders significant at .10, not included in model. Analysis of covariance modeled T2 BSS as function of arm & T1 BSS. Estimated mean difference in T2 scores calculated, no adjustment for multiple comparisons; Test type: Superiority; p = .07, ANCOVA; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-.29 to 8.0]
Statistical Analysis 2: Comparison: Waitlist Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .94, Regression, Linear; Mean Difference (Final Values) = -.01, 95% CI 2-sided [-3.3 to 3.1]
Statistical Analysis 3: Comparison: WtoH Intervention; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .06, one-sample t-test; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-7.0 to .12]

3. Secondary Outcome: Beck Depression Inventory (BDI -II)
Description: The Beck Depression Inventory-Second Edition (BDI-II) is a self-report instrument measuring the severity of common depressive symptoms. Each of its 21 items is rated on a 4-point Likert scale ranging from 0 to 3; total scores range from 0 to 63, with higher scores indicating greater degrees of depressive symptomatology. High levels of internal consistency (Cronbach α = 0.93) have been reported as well as concurrent validity with the BDI (r = 0.64 to r = 0.75), and the BHS among those with TBI (r = 0.60) (Beck and Steer, 1998) and general population samples (r = 0.52 to r = 0.63). (Beck and Steer, 1993). BDI-II outcome administered at the following study timepoints: Time 1 (Baseline for both arms), Time 2 (Post-Intervention for WtoH Intervention arm and Baseline 2 for Waitlist Control arm), and Time 3 Assessment (3 month follow up for WtoH Intervention arm and Post-Intervention for Waitlist Control arm
Time Frame: Time 2 BDI-II was assessed 3-months after Time 1 baseline assessment for both arms of the trial. Time 3 BDI-II was assessed 6 months after Time 1 baseline for both arms of the trial.
Population: n=14 WtoH and n=16 Waitlist BDI-II analyzed at Time 3 due to loss to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WtoH Intervention | Waitlist Control
Number analyzed (Participants) | 15 | 20
score on a scale
  Time 2 BDI-II | 26.8 (12.9) | 27.0 (9.4)
  Time 3 BDI-II: number analyzed (Participants) | 14 | 16
  Time 3 BDI-II | 24.9 (12.8) | 17.9 (12.0)
Statistical Analysis 1: Comparison: WtoH Intervention vs Waitlist Control; Analyses 2-sided test w/ sig level .05. N=35 analyzed w/ α .05 provided 80% power to detect effect size d=1. T1 variables compared using Wilcoxon rank sum & Fisher exact tests. Per protocol analysis, all participants required T2 BHS. T2 BDI compared bet arms controlling for T1 BDI. No confounders significant at .10, not included in model. Analysis of covariance modeled T2 BDI as function of arm & T1 BDI. Estimated mean difference in T2 scores calculated, no adjustment for multiple comparisons; Test type: Superiority; p = .13, ANCOVA; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-1.7 to 12.9]
Statistical Analysis 2: Comparison: Waitlist Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .003, Regression, Linear; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-13.8 to -3.6]
Statistical Analysis 3: Comparison: WtoH Intervention; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .002, one-sample t-test; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-18.0 to -5.3]

ADVERSE EVENTS:
Description: Definition does not differ from clinicaltrials.gov
Arm/Group | WtoH Intervention | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 0/15 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No